CLINICAL TRIAL: NCT02204007
Title: Comparison of Acetabular Shell Position Using 3D Planning vs. Standard Preoperative Planning: A Randomized Clinical Trial
Brief Title: Real Time 3D Imaging and Surrogate Bone Model
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Small number of subjects
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-555
Record Dates: First submitted 2014-07-28; First posted 2014-07-30 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-02

CONDITIONS: Arthritis
Keywords: Acetabular Shell; Total Hip Arthroplasty; 3D imaging
MeSH Terms: conditions — Arthritis | interventions — Imaging, Three-Dimensional

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 3D imaging, surrogate bone model (Experimental): 3D imaging & surrogate bone model
  Interventions: Device: 3D imaging & surrogate bone model
- Standard of Care Preoperative Imaging (No Intervention): Patients receiving standard of care preoperative planning prior to total hip arthroplasty.

INTERVENTIONS:
Device: 3D imaging & surrogate bone model — 3D imaging & surrogate bone model to assist with acetabular shell placement. Different that standard of care preoperative imaging
  Arms: 3D imaging, surrogate bone model

SUMMARY:
This is an observer-blinded prospective randomized clinical trial to define the efficacy of a new technology developed at the Cleveland Clinic to improve the positioning of the acetabular shell in total hip arthroplasty.The proposed study will enroll patients that have consented to total hip arthroplasty with or without screw fixation for treatment of hip pathology. This treatment is standard of care. Patients will receive standard of care pre- and post-operative care and placement of standard of care implants all of which are commercially available and FDA approved for general use for the clinical indications used in these patients. The only difference in treatment between the groups will be the use of a surrogate bone model to help assist the surgeon visualize the ideal placement of the acetabular component. Diagnostic testing performed specifically related to this study consists of obtaining one pre-operative and one post-operative CT scan. The post-operative scan is to be performed within two weeks of surgery.

The investigators predict that those patients with 3D imaging and bone model will have better acetabular shell placement than those with standard preoperative planning.

DETAILED DESCRIPTION:
The plan is enroll 44 subjects (22 in the standard surgery group and 22 in the experimental surgical group) into this randomized clinical trial. All subjects will have the standard of care indications for THA and will give informed consent for both the surgery and participation in this study. Enrollment will occur as part of the routine office evaluation and will be obtained by the treating surgeon or by the research assistant. Four surgeons (Wael Barsoum, Trevor Murray, Carlos Higuera, and Michael Bloomfield) with surgical experience in total hip arthroplasty will perform the procedures in this study. All subjects within each surgeon's practice who qualify for participation in this study will be approached. Subjects will be enrolled at least 10 days prior to the date of surgery. Ten days is the minimum time necessary to obtain a pre-operative CT scan for surgical planning and to manufacture the surrogate bone model. Patients who are not approached during regular office visits will be contacted by phone and if they are interested, they will be scheduled to arrive to the radiology department to sign the informed consent and receive the preoperative CT scan. Subjects will be randomized into either the experimental or control group at the time of consent by the study coordinator. Subjects in the experimental group will have their pre-operative planning done using the 3D surgical simulator and surrogate bone model will be available for the surgeon during surgery. Subjects in the control group will have their pre-operative planning done using plain film x-ray and two-dimensional (2D) templates.

Eligible subjects for inclusion in the study will be able to receive a pelvic CT scan at the Cleveland Clinic. Additionally, we will obtain standard of care pre- and post-operative x-rays (AP view). For subjects randomized into the experimental group, their CT scan DICOM images will be uploaded into the Cleveland Clinic developed surgical simulator specifically designed for THA at least 10 days prior to surgery. For each experimental subject, the Cleveland Clinic pre-operative planning software will be used to define the optimal size and location of the acetabular components (acetabular shell, and the ultra-high molecular weight polyethylene bearing - UHMWPE). The treating surgeon will virtually place the implant in the simulator software. The specification for shell placement will vary depending on the subject's individual pathology and pelvic morphology, but is expected to fall within the range of 10-35 degrees of anteversion and 30-50 degrees of abduction.

In the control group, each surgeon will use their standard methods of pre-operative planning using the pre-operative x-rays. To prepare the acetabulum and place the implants on the day of surgery, surgeons will use standard surgical alignment instruments provided by the manufacturer of the implant. For the experimental group, the surgeon will use CT scan and a 3D preoperative planning software to place the implants virtually. The surgeons are provided with a surrogate bone model with a fabricated acetabular implant placed in the same orientation as was planned in the surgical simulator software, and will use standard surgical instruments provided by the manufacturer of the implant.

The images obtained from the post-operative CT scans will be uploaded into the simulator software for 3D reconstruction. The 3D image of the post-operative pelvis with the implants will be superimposed onto the image of the pre-operative pelvis with the virtually placed implants. Using measurement tools within the software we will compare the position of the actual acetabular component placed in the patient with the desired position specified by the plan. The measurements that will be made are for angular orientations in 3D space (anteversion and inclination). Measurements are accurate to within a fraction of a degree.

ELIGIBILITY:
Inclusion Criteria:

* Subjects to be included in this protocol will be adult males and females of all races and socioeconomic status meeting the following criteria:
* Primary, unilateral Total hip arthroplasty (THA)
* 18 to 85 years old at time of surgery
* Able to get a pre- and post-operative CT scan at the Cleveland Clinic Main Campus at least 10 days prior to surgery

Exclusion Criteria:

* Significant metal in the joint that results in metal artifact on the pre--operative CT scan, thereby compromising the ability to visualize the acetabulum on the pre-operative simulator.
* Pregnancy
* Incarceration
* Condition deemed by physician or medical staff to be non-conducive to patient's ability to complete the study, or a potential risk to the patient's health and well-being.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Higuera, MD, Principal Investigator — The Cleveland Clinic; Alison Klika, MS, Study Director — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Codsi MJ, Bennetts C, Gordiev K, Boeck DM, Kwon Y, Brems J, Powell K, Iannotti JP. Normal glenoid vault anatomy and validation of a novel glenoid implant shape. J Shoulder Elbow Surg. 2008 May-Jun;17(3):471-8. doi: 10.1016/j.jse.2007.08.010. Epub 2008 Mar 7. PMID 18328741
- [Background] Scalise JJ, Bryan J, Polster J, Brems JJ, Iannotti JP. Quantitative analysis of glenoid bone loss in osteoarthritis using three-dimensional computed tomography scans. J Shoulder Elbow Surg. 2008 Mar-Apr;17(2):328-35. doi: 10.1016/j.jse.2007.07.013. Epub 2008 Jan 22. PMID 18218326
- [Background] Scalise JJ, Codsi MJ, Bryan J, Iannotti JP. The three-dimensional glenoid vault model can estimate normal glenoid version in osteoarthritis. J Shoulder Elbow Surg. 2008 May-Jun;17(3):487-91. doi: 10.1016/j.jse.2007.09.006. Epub 2008 Feb 20. PMID 18282721
- [Background] Scalise JJ, Codsi MJ, Bryan J, Brems JJ, Iannotti JP. The influence of three-dimensional computed tomography images of the shoulder in preoperative planning for total shoulder arthroplasty. J Bone Joint Surg Am. 2008 Nov;90(11):2438-45. doi: 10.2106/JBJS.G.01341. PMID 18978413
- [Background] Eisler T, Svensson O, Tengstrom A, Elmstedt E. Patient expectation and satisfaction in revision total hip arthroplasty. J Arthroplasty. 2002 Jun;17(4):457-62. doi: 10.1054/arth.2002.31245. PMID 12066276
- [Background] Furnes O, Lie SA, Espehaug B, Vollset SE, Engesaeter LB, Havelin LI. Hip disease and the prognosis of total hip replacements. A review of 53,698 primary total hip replacements reported to the Norwegian Arthroplasty Register 1987-99. J Bone Joint Surg Br. 2001 May;83(4):579-86. doi: 10.1302/0301-620x.83b4.11223. PMID 11380136
- [Background] Older J. Charnley low-friction arthroplasty: a worldwide retrospective review at 15 to 20 years. J Arthroplasty. 2002 Sep;17(6):675-80. doi: 10.1054/arth.2002.31973. PMID 12216018
- [Background] Phillips CB, Barrett JA, Losina E, Mahomed NN, Lingard EA, Guadagnoli E, Baron JA, Harris WH, Poss R, Katz JN. Incidence rates of dislocation, pulmonary embolism, and deep infection during the first six months after elective total hip replacement. J Bone Joint Surg Am. 2003 Jan;85(1):20-6. doi: 10.2106/00004623-200301000-00004. PMID 12533567
- [Background] Parvizi J, Wade FA, Rapuri V, Springer BD, Berry DJ, Hozack WJ. Revision hip arthroplasty for late instability secondary to polyethylene wear. Clin Orthop Relat Res. 2006 Jun;447:66-9. doi: 10.1097/01.blo.0000218751.14989.a6. PMID 16672896
- [Background] Alberton GM, High WA, Morrey BF. Dislocation after revision total hip arthroplasty : an analysis of risk factors and treatment options. J Bone Joint Surg Am. 2002 Oct;84(10):1788-92. PMID 12377909
- [Background] Dorr LD, Wolf AW, Chandler R, Conaty JP. Classification and treatment of dislocations of total hip arthroplasty. Clin Orthop Relat Res. 1983 Mar;(173):151-8. PMID 6825326
- [Background] McCollum DE, Gray WJ. Dislocation after total hip arthroplasty. Causes and prevention. Clin Orthop Relat Res. 1990 Dec;(261):159-70. PMID 2245542
- [Background] Robinson RP, Simonian PT, Gradisar IM, Ching RP. Joint motion and surface contact area related to component position in total hip arthroplasty. J Bone Joint Surg Br. 1997 Jan;79(1):140-6. doi: 10.1302/0301-620x.79b1.6842. PMID 9020463
- [Background] Mahomed NN, Barrett JA, Katz JN, Phillips CB, Losina E, Lew RA, Guadagnoli E, Harris WH, Poss R, Baron JA. Rates and outcomes of primary and revision total hip replacement in the United States medicare population. J Bone Joint Surg Am. 2003 Jan;85(1):27-32. doi: 10.2106/00004623-200301000-00005. PMID 12533568
- [Background] Hafez MA, Chelule KL, Seedhom BB, Sherman KP. Computer-assisted total knee arthroplasty using patient-specific templating. Clin Orthop Relat Res. 2006 Mar;444:184-92. doi: 10.1097/01.blo.0000201148.06454.ef. PMID 16446589
- See also: Medical Device Materials — http://www.dsm.com/markets/medical/en_US/home.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 3D Imaging, Surrogate Bone Model | Standard of Care Preoperative Imaging
Started | 18 | 18
Completed | 17 | 17
Not Completed | 1 | 1
Not completed — Surgery Canceled | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3D Imaging, Surrogate Bone Model | Standard of Care Preoperative Imaging | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Continuous [Mean (Full Range); unit: years] | 65.4 [44 to 80] | 58.6 [41 to 82] | 62.0 [41 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 14
  Male | 8 | 12 | 20

OUTCOME MEASURES:

1. Primary Outcome: Acetabular Shell Version and Inclination
Description: A CT scan of all patients will be obtained within 2 weeks of surgery to measure placement (acetabular version & inclination measured in degrees) of the acetabular shell
Time Frame: within 2 weeks of surgery
Measure: Mean (Full Range); unit: degrees
Arm/Group | 3D Imaging, Surrogate Bone Model | Standard of Care Preoperative Imaging
Number analyzed (Participants) | 14 | 11
degrees
  Inclination | 43.4 [34 to 54] | 39.3 [27 to 55]
  Anteversion | 27.1 [9 to 48] | 23.3 [9 to 37]

2. Secondary Outcome: Operative Time
Description: Duration of the surgical case
Time Frame: time of surgery
Measure: Mean (Full Range); unit: minutes
Arm/Group | 3D Imaging, Surrogate Bone Model | Standard of Care Preoperative Imaging
Number analyzed (Participants) | 14 | 11
minutes | 128.9 [76 to 179] | 151.2 [82 to 291]

ADVERSE EVENTS:
Arm/Group | 3D Imaging, Surrogate Bone Model | Standard of Care Preoperative Imaging
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No